CLINICAL TRIAL: NCT01691040
Title: Phase IIa Study to Characterize the Effects of the Spiegelmer® NOX H94 on Anemia of Chronic Disease in Patients With Cancer
Brief Title: Efficacy of NOX-H94 on Anemia of Chronic Disease in Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNOXH94C201; 2012-001525-27 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2012-09-24 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Anemia of Chronic Disease
Keywords: Hepcidin; Iron; Anemia of Chronic Disease; Anemia; Cancer; Interleukin-6; Iron restriction; Lymphoma; CLL; Multiple Myeloma; Hodgkin; anti-hepcidin
MeSH Terms: conditions — Anemia; Neoplasms; Lymphoma; Multiple Myeloma | interventions — NOX-H94

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label pilot group (Experimental): Twice weekly administration of NOX-H94
  Interventions: Drug: NOX-H94; Drug: Placebo solution

INTERVENTIONS:
Drug: NOX-H94 — intravenous injection
  Other Names: lexaptepid pegol
Drug: Placebo solution — intravenous injection
  Other Names: Glucose 5%

SUMMARY:
This study is conducted to determine the safety, tolerability, and efficacy of NOX-H94 in patients with anemia of chronic disease (ACD). Furthermore, this study is intended to provide data needed to correlate plasma concentrations of NOX-H94 with its efficacy and to choose the appropriate dose and dose schedule of subsequent efficacy studies.

Some chronic diseases, e.g. tumors, inflammation, renal disease, are associated with high hepcidin concentrations in the blood. These hepcidin concentrations cause a reduction in iron concentrations in the blood and subsequently impair formation of red blood cells. Treatment with NOX-H94 is expected to inhibit this patho-mechanism by binding and inactivating hepcidin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Female or male aged >18 years
* Clinically significant anemia of chronic disease (ACD) attributed to histologically or cytologically proven malignancy, either hematological or solid tumor, of any grade or stage: Hemoglobin (Hb) 7.0 g/dL to 10 g/dL, Transferrin saturation (TSAT) <50%, Serum iron <50 µg/dL (SI: <9.0 µmol/L), AND Ferritin >30 ng/mL (SI: >30 µg/L)
* Previous treatment with systemic anti-cancer therapy / regimen
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Estimated life expectancy ≥12 weeks
* Men must agree to follow effective contraception methods during treatment and for 3 months after completion of treatment. Women of childbearing potential must agree to use two forms of effective contraception during treatment and for 3 months after completion of treatment.

Exclusion Criteria:

* Inability to personally provide written informed consent or to understand and collaborate throughout the study
* History of pure red cell aplasia, thalassemia major or sickle cell disease History of anemia unrelated to cancer <10 g/dL within 6 months prior to screening
* Uncorrected iron deficiency
* Regular need for blood transfusions at intervals <6 weeks
* Acute or myeloid leukemia
* Known or suspected chronic bleeding
* Tumor with gastro-intestinal involvement without negative test for fecal occult blood
* Suspected or known history of hemochromatosis
* Known infection with human immunodeficiency virus, hepatitis B, or hepatitis C
* Impaired liver function with bilirubin ≥2.0 mg/dL (26 μmol/L), AST or ALT ≥2 times upper limit
* History or risk of significant hepatic disease, e.g. chronic alcohol abuse, hepatic steatosis, hepatic cirrhosis, or organ transplantation
* Severe renal impairment: estimated glomerular filtration rate (eGFR) <30 mL/min (Cockcroft-Gault)
* Known central nervous system malignancy or metastasis
* Significant cardiac disease (e.g. uncontrolled hypertension: systolic blood pressure [BP] >150 mmHg or diastolic BP >100 mmHg; myocardial infarction or unstable angina pectoris) within 6 months prior to screening
* Positive pregnancy test (serum ß-hCG at screening, urine pregnancy test prior to first treatment) or lactation
* Previous participation in this study or treatment with an investigational agent <21 days prior to treatment start
* Hemolysis or bleeding >500 mL (measured or estimated) within 6 weeks prior to treatment start
* Treatment with erythropoiesis-stimulating agents (ESAs) or red blood cell (RBC) transfusions <21 days prior to treatment start
* Cytotoxic anti-tumor treatment <21 days prior to treatment start or planned during the anticipated study period (within 3 months from treatment start or randomization). Maintenance therapy is permitted throughout the study (e.g. lenalidomide, interferon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Response rate of anemia | treatment start to 1 week after treatment end
  • Hb increase ≥1 g/dL OR reticulocyte index normalization (≥1%) at any time point until 1 week after the end of treatment
  AND absence of all of the following treatment failure criteria until 1 week after the end of treatment:
  * Erythrocyte transfusion, ESA or IV iron,
  * Hb drop by ≥1 g/dL
  * Treatment interruption due to adverse events (AEs)

SECONDARY OUTCOMES:
Response | Treatment start to 8 weeks after end of treatment
  Proportion of treatment responders at study visits V4, V6, V8, and V10 to V14, as defined for the primary efficacy endpoint
Failure | Treatment start to 1 week after end of treatment
  Proportion of treatment failures at study visits V4, V6, V8, and V10, as defined for the primary efficacy endpoint
Safety and tolerability | Treatment start to 8 weeks after end of treatment
  Adverse events, Safety signals derived from laboratory diagnostics, vital signs.
Pharmacokinetics | Treatment start to 8 weeks after end of treatment
  NOX-H94 plasma concentrations
Reticulocytes | Treatment start until 8 weeks after end of treatment
  Absolute values and change from baseline
Red blood cells | Treatment start until 8 weeks after end of treatment
  Absolute values and change from baseline
Transferrin | Treatment start to 8 weeks after end of treatment
  Absolute concentrations and change from baseline
Serum iron | Treatment start to 8 weeks after end of treatment
  Absolute concentrations and change from baseline
Ferritin | Treatment start to 8 weeks after end of treatment
  Absolute concentrations and change from baseline
Transferrin saturation | Treatment start to 8 weeks after end of treatment
  Absolute concentrations and change from baseline
Hemoglobin | Treatment start to 8 weeks after end of treatment
  Absolute concentrations and change from baseline

OTHER OUTCOMES:
Exploratory analyses | Treatment start to 1 week after end of treatment
  Soluble transferrin receptor
Exploratory analyses | Treatment start to 1 week after end of treatment
  Reticulocyte hemoglobin content

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — TME Pharma AG
Locations (11):
- Austria (3):
  - University Hospital, Graz
  - AKH Vienna, Vienna
  - Wilhelminenspital, Vienna
- Bulgaria (3):
  - University Hospital, Plovdiv
  - Tokuda Hospital, Sofia
  - University Hospital, Varna
- Romania (5):
  - Spitalul Judetean, Brasov
  - Institutul Oncologic, Cluj-Napoca
  - Spitalul Municipal, Craiova
  - Spitalul Judetean, Târgu Mureş
  - Oncomed, Timișoara

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581